CLINICAL TRIAL: NCT04951180
Title: Arthroscopic Treatment for Femoral Acetabular Impingement Syndrome With Gluteus Medius Lesions.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: M2021221
Record Dates: First submitted 2021-06-27; First posted 2021-07-06 (Actual); Last update posted 2021-07-07 (Actual); Status verified 2021-06

CONDITIONS: Femoral Acetabular Impingement
MeSH Terms: conditions — Femoracetabular Impingement | interventions — Demography

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Group 1: Femoral acetabular impingement syndrome (FAIS) patients with gluteus medius lesions
  Interventions: Other: Demographic data and MRI images extraction

INTERVENTIONS:
Other: Demographic data and MRI images extraction — The data were retrospectively extracted pre- and postoperatively after hip arthroscopy. The prognosis of the surgery was evaluated through MRI images.

SUMMARY:
To evaluate the prognosis of femoral acetabular impingement syndrome (FAIS) patients with gluteus medius lesions after hip arthroscopy.

DETAILED DESCRIPTION:
The data of FAIS patients with gluteus medius lesions were retrospectively extracted pre- and postoperatively after hip arthroscopy. The prognosis of the surgery was evaluated through MRI images.

ELIGIBILITY:
Inclusion Criteria

* Diagnosed FAIS
* Ineffective conservative treatment
* Available pre- and postoperative images

Exclusion Criteria

* Revision arthroscopy
* Osteoarthritis
* History of hip joint disease or surgery
* Sacroiliac joint disease
* Loss of follow-up

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Femoral acetabular impingement syndrome (FAIS) patients with gluteus medius lesions.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2021-05-01 (Actual); Primary Completion 2021-08-01 (Estimated); Study Completion 2021-12-01 (Estimated)

PRIMARY OUTCOMES:
MRI images | at least 1-year after hip arthroscopy
  Characteristics of postoperative MRI images

CONTACTS AND LOCATIONS:
Overall Officials: Jian-quan Wang, M.D., Study Chair — Peking University Third Hospital
Locations (1):
- Peking University Third Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No